CLINICAL TRIAL: NCT02811445
Title: Role of the Gut Microbiome and Serum Metabolome on Lean Mass and Physical Function in Older Adults
Brief Title: Role of the Gut Microbiome on Lean Mass and Physical Function in Older Adults
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Michael, Scientist II, Tufts University
Other Study IDs: GRANT11960287
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Sarcopenia
Keywords: microbiome, metabolome, aging, lean mass, physical function
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Feces, Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High Functioning: Defined by a short physical performance battery score (SPPB) greater than or equal to 11.
- Low Functioning: Defined by a short physical performance battery score (SPPB) less than or equal to 7.

SUMMARY:
The investigators recently published significant associations between circulating gut bacteria-related metabolites with lean and skeletal muscle mass and with measures of physical function in older adults, evidence that suggests a role for gut bacteria on the maintenance of these outcomes. To date, studies aimed at identification of associations between gut bacteria with lean mass or with specific measures of physical function have yet to be reported. Accordingly, the over-arching hypothesis is that gut bacteria are associated with, and are causatively involved in mechanisms that underlie the maintenance of lean mass and physical function in older adults. Results obtained from the proposed study are intended as the basis for future studies aimed at targeted modulation of the gut microflora, which may be a novel and innovative means for improving lean mass and physical function, and for addressing the public health priority of healthy aging in older adults.

DETAILED DESCRIPTION:
In older adults (70+ years), reduced lean body mass and physical function are associated with increased disability, hospitalization, morbidity and mortality. Because older adults are the fastest growing global subpopulation, identification of mechanisms that underlie the maintenance of lean mass and physical function will be important for addressing the public health priority of healthy aging.

Gut bacteria may be involved in mechanisms that underlie the maintenance of lean mass and physical function. In support of this hypothesis, in multiple publications the investigators recently reported significant associations between circulating gut bacteria-related metabolites with these outcomes in older adults. Accordingly, the overarching study hypothesis is that is gut bacteria are associated with, and are causatively involved in mechanisms that underlie the maintenance of lean mass and physical function in older adults. To test this hypothesis, the investigators propose to: characterize the association between fecal bacteria with lean mass and physical function (AIM 1), test the causative role of gut bacteria on the maintenance of lean mass and physical function by colonizing germ-free mice with fecal bacteria from older adults (AIM 2), and examine potential mechanisms that link gut bacteria with these outcomes by identifying associations between gut bacteria and serum metabolites with lean mass and physical function (AIM 3).

ELIGIBILITY:
Inclusion Criteria:

i) Willing and able to sign the IRB approved informed consent form ii) Male and Female iii) 70-85 years of age iv) BMI ≤ 35 kg/m2 v) Willing to come to the HNRCA laboratory for baseline and 1-month follow-up study visits vi) SPPB ≥ 11 ("High-Functioning", HF; 20 subjects: 10 males, 10 females) vii) 4 ≤ SPPB ≤ 7 ("Low-Functioning", LF; 20 subjects: 10 males, 10 females)

Exclusion Criteria:

i) Non-English speaker ii) Acute or terminal illness iii) Surgery in the past 6 months iv) Lower extremity fracture within the past 6 months v) Myocardial infarction in the past 6 months vi) Coronary artery disease, peripheral vascular disease, previous stroke, or history of transient ischemic attacks vii) Cognitive impairment (MMSE score < 23) viii) Uncontrolled hypertension (> 160/100 mmHg) ix) Neuromuscular disease or drugs affecting neuromuscular function x) Androgen therapy in males xi) Estrogen therapy in females xii) Significant immune disorder xiii) Kidney Failure xiv) Pancreatic disease xv) Diabetes xvi) Gastrointestinal or malabsorption diseases xvii) History of cholecystectomy xviii) Use of probiotics, prebiotics or antibiotics in the past 3 months xix) The subject has any other condition, which in the opinion of the Investigator, precludes the subject's participation in the trial.

xx) With the goal of matching the HF and LF groups for age, sex,and BMI, subjects may be excluded because their age, sex or BMI puts them outside the range needed for this study.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults (70-85y), BMI < 35 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S lustgarten, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: 5/2016 to 2/2018 at the Tufts University Human Nutrition Research Center on Aging (Boston, MA). Sedentary older adults were recruited from a database of older adults, and via advertisements posted on HNRCA bulletin boards and online media.
Pre-assignment Details: Exclusion criteria included a SPPB score of 9 or 10, a BMI ≥ 35 kg/m2, acute or terminal illness, myocardial infarction in the past 6 months, unstable cardiovascular disease, MMSE score < 23, blood pressure > 150/90 mm Hg, androgen therapy in males, estrogen therapy in females, and others.
Period: Overall Study
Arm/Group | High Functioning | Low Functioning
Started | 18 | 11
Completed | 18 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Functioning | Low Functioning | Total
Number analyzed (Participants) | 18 | 11 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.9 (3.42) | 77.0 (4.43) | 76.3 (3.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 10 | 6 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 11 | 29
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (3.5) | 27.6 (3.7) | 28.0 (3.6)
Percentage of whole body lean mass [Mean (Standard Deviation); unit: Percentage of whole body mass] — Higher values for the percentage of whole body lean mass are indicative of a better body composition, when compared with lower values.
  Percentage of whole body mass | 67.3 (6.4) | 62.2 (6.4) | 65.7 (6.6)
Short physical performance score (SPPB) [Mean (Standard Deviation); unit: scores on a scale] — The Short Physical Performance Score (SPPB) is a combined measure of physical function that includes balance, a chair stand test (the time required to complete 5 chair stands), and the time needed to walk 4 meters. Each of these 3 tests are scored from 0 to 4. The scores for each individual test are summed, and accordingly, the lowest possible SPPB score would be 0, and the highest would be 12. A score of 12 would indicate good physical function, whereas a score of 0 is indicative of poor physical function.
  scores on a scale | 11.5 (0.74) | 7.64 (1.29) | 10.1 (2.2)
400-meter gait speed [Mean (Standard Deviation); unit: meters/second] — The 400-meter gait speed test measures the time needed to walk 400 meters. A shorter time is indicative of good physical function, whereas a longer time indicates worse physical function.
  meters/second | 1.13 (0.16) | 0.96 (0.16) | 1.10 (0.18)
Leg press 1 repetition maximum value [Mean (Standard Deviation); unit: Newtons] — The leg press one repetition value represents the maximum amount of the weight that the participant was able to push with their legs. A higher value is indicative of higher muscle strength, whereas lower values indicate lower muscle strength.
  Newtons | 1878 (677) | 1407 (535) | 1699 (653)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Whole Body Lean Mass (%WBLM)
Description: %WBLM measured with dual x-ray absorptiometry (DXA). A higher %WBLM is indicative of a higher amount of whole-body lean mass, when compared with lower values.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: % of whole body mass
Arm/Group | High Functioning | Low Functioning
Number analyzed (Participants) | 18 | 11
% of whole body mass | 67.3 (6.77) | 61.9 (6.64)

2. Primary Outcome: Physical Function Measurement
Description: Short physical performance battery (SPPB) score. The SPPB is a combined measure of physical function that includes balance, a chair stand test (the time required to complete 5 chair stands), and the time needed to walk 4 meters. Each of these 3 tests are scored from 0 to 4. The scores for each individual test are summed, and accordingly, the lowest possible SPPB score would be 0, and the highest would be 12. A score of 12 would indicate good physical function, whereas a score of 0 is indicative of poor physical function.
Time Frame: 1-month
Measure: Mean (Standard Deviation); unit: score
Arm/Group | High Functioning | Low Functioning
Number analyzed (Participants) | 18 | 11
score | 11.2 (1.1) | 7.4 (1.5)

3. Primary Outcome: 400-meter Gait Speed
Description: Measurement of 400-meter gait speed at the 1-month study visit compared against baseline. A slower time to walk 400 meters is indicative of worse physical function, when compared with a faster time.
Time Frame: 1-month
Measure: Mean (Standard Error); unit: meters/second
Arm/Group | High Functioning | Low Functioning
Number analyzed (Participants) | 18 | 11
meters/second | 1.12 (0.16) | 0.96 (0.19)

4. Primary Outcome: Leg Press 1 Repetition Maximum
Description: Measurement of the leg press 1 repetition maximum at the 1-month study visit compared with baseline. The leg press 1 repetition maximum test involves the maximum amount of weight that the participant can push with their legs. A higher value is indicative of higher muscle strength, when compared with lower values.
Time Frame: 1-month
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | High Functioning | Low Functioning
Number analyzed (Participants) | 18 | 11
Newtons | 1863.9 (665.1) | 1343.2 (565.3)

ADVERSE EVENTS:
Time Frame: Study participants were observed at two time points that were one month apart (baseline and a 1-month study visit).
Arm/Group | High Functioning | Low Functioning
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/11
Other Adverse Events (participants affected / at risk) | 0/18 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT02811445/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT02811445/SAP_001.pdf